CLINICAL TRIAL: NCT01321034
Title: Effect of Niacin in the Lipoprotein (a) Concentration With Regard to Apolipoprotein (a) Size and Baseline Lipoprotein (a) Concentration.
Brief Title: Effect of Niacin in the Lipoprotein (a) Concentration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Aragones de Ciencias de la Salud (Other Government)
Collaborators: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Fernando Civeira, Chief Lipid Clinic. Hospital Universitario Miguel Servet de Zaragoza, Spain, Instituto Aragones de Ciencias de la Salud
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2010-022258-17
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Hypercholesterolemia
Keywords: Lipoprotein (a); LPA; Niacin; Kringle IV-2 repeats
MeSH Terms: conditions — Hypercholesterolemia | interventions — Niacin; MK-0524

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Niacin/Laropiprant (Other): Subjects with normal Lp(a) will be use as comparative group for the other two groups, so no placebo group is required is this study
  Interventions: Drug: Niacin/Laropiprant

INTERVENTIONS:
Drug: Niacin/Laropiprant — 1g/20 mg day of Niacin/Laropiprant for 4-weeks followed by 8 additional weeks of 2 g/40 mg day.

SUMMARY:
Objectives.

* To evaluate the absolute and relative Lp(a) lowering effect of 1g/20 mg and 2 g/40 mg day of Niacin/Laropiprant in subjects with normal Lp(a) (< 30 mg/dL), high Lp(a) (30-60 mg/dL) and very high Lp(a) (> 60 mg/dL).
* To evaluate the absolute and relative Lp(a) lowering effect of 1g/20 mg and 2 g/40 mg day of Niacin/Laropiprant depending on the number of kringle IV-2 repeated copies on the apo(a) gene. 2.1.1 Hypotheses.
* The Lp(a) lowering effect of niacin is dependent of the pre-treatment Lp(a) concentration, with higher absolute and relative reduction in Lp(a) in subjects with hyperlipoproteinemia(a).
* Lp(a) size, throughout modifying hepatic synthesis of apo(a), is a major factor related to the lowering effect variability of niacin in human.

DETAILED DESCRIPTION:
Open-label 12-week study, 1g/20 mg day of Niacin/Laropiprant for 4-weeks followed by 8 additional weeks of 2 g/40 mg day. Subjects with normal Lp(a) will be use as comparative group for the other two groups, so no placebo group is required is this study.

Subjects: volunteers from the Lipid Clinic of Hospital Universitario Miguel Servet of Zaragoza, Spain. Subjects were selected according to their previously determined Lp(a)concentration. All volunteers before any study procedure will have to give written inform consent to a protocol previously approved for the Ethical Committees of our institutions.

Biochemical determinations: lipids: total cholesterol and triglycerides; lipoproteins: HDL-cholesterol, Lp(a); apolipoproteins: Apo A1 and apo B and safety biochemical parameters (glucose, uric acid, creatinine, liver and muscle enzymes will be measured at baseline and at the end of the two treatment periods (weeks 4 and 8).

An adverse experience questionnaire will be done in each visit. Genetic analysis: apo(a) genetic polymorphism responsible of the Lp(a) size variability will be analyzed by a PCR-based methodology (Lanktree et al. J Lipid Res 2009; 50: 768-72 ).

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 and < 80 years
2. LDL cholesterol between 70 and 190 mg/dL
3. Triglycerides < 500 mg/dL
4. At least 2 Lp(a) determinations previous to the beginning of the study without differences >20% or > 20 mg/dL.
5. No lipid lowering therapy or on stable doses in the last 3 months

Exclusion Criteria:

1. Liver disease or liver enzymes >2 times higher than reference values
2. Creatinine > 2 mg/dL
3. Active peptic ulcer
4. Clinical gout in the last year
5. Uncontrolled diabetes (HbA1c >8%)
6. Enrolment in other drug clinical trial in the previous 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
absolute and relative Lp(a) lowering effect of 1g/20 mg and 2 g/40 mg day of Niacin/Laropiprant in subjects with normal Lp(a) (<30 mg/dL), high Lp(a) (30-60 mg/dL) and very high Lp(a) (>60 mg/dL g/40 mg day of Niacin/Laropiprant | 8 weeks

SECONDARY OUTCOMES:
absolute and relative Lp(a) lowering effect of 1g/20 mg and 2 g/40 mg day of Niacin/Laropiprant depending on the number of kringle IV-2 repeated copies on the apo(a) gene. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Civeira, MD, Principal Investigator — Hospital Miguel Servet
Locations (3):
- Spain (3):
  - Hospital San Jorge, Huesca
  - Hospital Universitario Miguel Servet, Zaragoza
  - Hospital Royo Villanova, Zaragoza